CLINICAL TRIAL: NCT00802802
Title: Dose-Finding and Pharmacogenetic Study of Efavirenz in HIV-infected and HIV/TB Co-infected Infants and Children 3 Months to Less Than 36 Months of Age
Brief Title: Efavirenz (EFV) in HIV-Infected and HIV/Tuberculosis (TB) Coinfected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1070; 10633 (Registry Identifier: DAIDS ES); IMPAACT P1070
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — efavirenz

ARMS (3):
- Cohort I, Step 1 (Experimental): HIV-infected children 3 months to 36 months of age, receiving EFV and two NRTIs
  Interventions: Drug: Efavirenz (EFV)
- Cohort II (Experimental): HIV/TB-coinfected children 3 months to 36 months of age, receiving EFV, two NRTIs, and rifampin-containing anti-tuberculosis (anti-TB) therapy
  Interventions: Drug: Efavirenz (EFV); Drug: Rifampin-containing anti-TB therapy
- Cohort I, Step 2 (Experimental): HIV-infected children from Cohort I who become coinfected with TB during the study. They will receive EFV, two NRTIs, and rifampin-containing anti-TB therapy
  Interventions: Drug: Efavirenz (EFV); Drug: Rifampin-containing anti-TB therapy

INTERVENTIONS:
Drug: Efavirenz (EFV) — Participants will be administered oral EFV at a dose ranging from 50 mg to 800 mg once daily, based on weight and CYP 2B6 genotype. EFV capsules will be opened into a small amount of a compatible food or liquid vehicle; the smallest amount of food or liquid that will enable the child to swallow the capsule contents should be used (i.e., EFV should not be taken with a meal).
  Other Names: EFV
Drug: Rifampin-containing anti-TB therapy — Treatment with rifampin-containing anti-TB treatment regimen. Treatment will last at least 24 weeks and up to 36 weeks.
  Arms: Cohort I, Step 2; Cohort II

SUMMARY:
Efavirenz (EFV) is an anti-HIV medicine that is commonly used to treat HIV infection in adults and children older than 3 years of age. This study is being conducted to look at the safety of EFV, blood levels of EFV, genetic factors that may affect blood levels of EFV, and how easy it is for infants and young children to take and tolerate EFV. This information will help recommend the best doses of EFV for children younger than 3 years of age.

DETAILED DESCRIPTION:
An increasing number of children in resource-limited countries require treatment for both HIV and tuberculosis (TB); however, the options for antiretroviral therapy (ART) that is compatible with concurrent rifampin-containing anti-TB therapy are limited. As a result, treatment of HIV/TB-coinfected patients remains difficult with multiple drug interactions, very high pill burdens, overlapping toxicities, and possible immune reconstitution affecting treatment outcomes.

The use of EFV in adults and older children has allowed them to maintain their non-nucleoside reverse transcriptase inhibitor (NNRTI) backbone while receiving TB therapy including rifampin. In younger children with TB/HIV coinfection, the first-line treatment recommendation has been the triple-nucleoside reverse transcriptase inhibitor (NRTI) regimen. However, this regimen has been shown to be less effective than an EFV plus NNRTI-based regimen. In addition, triple-NRTI regimens in resource-limited settings are costly and have limited data in patients with TB, and monitoring for drug-related hypersensitivity reactions is difficult. All of these factors make EFV an attractive agent for use in HIV-infected pediatric patients with and without TB coinfection. This study will evaluate the safety, tolerance, and pharmacokinetics (PKs) of EFV when administered as opened capsules to pediatric patients younger than 3 years of age, with and without concomitant rifampin-containing anti-TB therapy. This study will also investigate genetic polymorphisms, including CYP 2B6, to help establish dosing guidelines.

This study will have two cohorts that will enroll at the same time. Cohort I, Step 1 will enroll HIV-infected infants without TB coinfection who are eligible for initiation of ART. Cohort I, Step 1 will be administered EFV for up to 24 weeks. EFV dosage, in Cohort I, Step 1, will range from 50 mg to 600 mg once daily, based on weight and CYP 2B6 genotype.

Participants in Cohort I Step 1 who develop TB or TB immune reconstitution inflammatory syndrome (IRIS) and require anti-TB medications will be allowed to enroll into Cohort I, Step 2, in which they will receive rifampin-containing anti-TB therapy and a higher dose of EFV (50 mg to 800 mg) to account for the anticipated impact of rifampin on EFV PKs. If participants in Cohort I, Step 2 require more than 24 weeks of anti-TB therapy and are unable to obtain EFV capsules from in-country sources, they may remain on the study longer than 24 weeks until discontinuing anti-TB therapy, up to 36 weeks study duration.

Participants in Cohort II will be HIV/TB coinfected infants who are eligible for ART and have been treated with and tolerated a rifampin-containing anti-TB treatment regimen for at least 1 week prior to enrollment. Participants in Cohort II will be followed while taking both rifampin-containing anti-TB and EFV therapy for 24 weeks; participants unable to obtain EFV capsules from in-country sources at the conclusion of the study may remain on the study until discontinuing anti-TB therapy, up to 36 weeks study duration. An estimated 10 to 20 of these participants from Cohort II will be followed every 4 weeks on study and provided EFV until completion of TB treatment (for up to 36 weeks study duration).

Participants in both cohorts will be stratified based on age. One stratification will include children 3 months to younger than 24 months of age, and the second stratification will include children 24 months to younger than 36 months of age. Participants will then be further stratified by cytochrome P450 genotype polymorphisms, including CYP 2B6. All participants will receive an EFV-based ART regimen using the capsule formulation of EFV and two NRTIs (chosen by site investigator). EFV capsules will be opened into a small amount of compatible, familiar, and locally available food or liquid (e.g., formula, expressed breast milk, mashed banana).

Study visits will occur at screening, entry, and at Weeks 2, 4, 6, 8, 12, 16, 20, and 24; some participants may continue to have a visit every 4 weeks after Week 24 until Week 36. At most visits, participants will undergo a physical exam, give a medical history, and have blood and urine collected. At some visits, dried blood spots (DBS) will be prepared and plasma samples will be stored. The Week 2 visit will also consist of intensive PK samplings where blood will be collected prior to taking the EFV dose and at 2, 4, 8, 12, and 24 hours post-dose. Individual dose adjustments may be made based on the results from the Week 2 visit.

ELIGIBILITY:
Inclusion Criteria (Cohort I, Step 1 and Cohort II)

* Older than 3 months but younger than 36 months of age (up to but not including the 3rd birthday) at the time of enrollment
* Documentation of HIV-1 infection defined as positive results from two samples collected at different time points. More details on this criterion can be found in the protocol.
* Treatment-eligible as defined by country-specific guidelines, World Health Organization (WHO) treatment algorithm, or by clinician's determination that the participant should be treated on other clinical grounds and will initiate antiretroviral (ARV) therapy (ART) AND has determined that in-country access to ART will be available at study conclusion
* Able to swallow the contents of efavirenz (EFV) as opened capsules in food or liquid vehicle
* Parent, legal guardian, or designated guardian according to country-specific guidelines able and willing to provide signed informed consent and to have the participant followed at the clinical site

Inclusion Criteria (Cohort I, Step 2 ONLY)

* Currently enrolled in Cohort I, Step 1
* Clinically diagnosed with HIV/TB co-infection and requires rifampin-containing therapy, in the clinical judgment of the site investigator
* Chemistry and hematology laboratory values drawn during Cohort I, Step 1 are all Grade 3 or lower, except for aspartate aminotransferase/alanine aminotransferase (AST/ALT), which must be Grade 2 or lower within 4 weeks of entry into Cohort I, Step 2

Inclusion Criteria (Cohort II ONLY)

* Clinically diagnosed with HIV/TB coinfection and requires rifampin-containing therapy, in the clinical judgment of the site investigator
* Participant is tolerating a rifampin-containing anti-TB drug regimen for at least 1 week prior to study entry
* Participant plans to continue anti-TB and study treatment for at least 16 weeks from initiation of study treatment

Exclusion Criteria (Cohort I, Step 1 and Cohort II)

* Known hypersensitivity to any component of EFV capsule formulation.
* Participants with severe malnutrition defined in the protocol
* Infants/children who have previously been treated with EFV-based ART
* Infants/children younger than 24 months of age with documented receipt of nevirapine (NVP) therapy, including single dose NVP for prevention of mother-to-child transmission (PMTCT). More information on this criterion can be found in the protocol.
* Infants/children younger than 24 months of age whose mothers have documentation of receiving NVP as part of PMTCT unless they meet criteria under the exception detailed in the protocol. More information on this criterion can be found in the protocol.
* Grade 2 or higher AST or ALT at screening
* Any Grade 3 or higher laboratory toxicity at screening
* Higher than Grade 3 clinical toxicity at screening
* Participants with acute, serious infections requiring active treatment (e.g. pneumocystis pneumonia [PCP], etc.) may not enroll until judged to be clinically stable by the site investigator. Participants may enroll while completing active opportunistic infection treatment. Prophylaxis against opportunistic infections, including isoniazid, will be allowed.
* Chemotherapy for active malignancy
* Active central nervous system (CNS) infection, such as TB meningitis or cryptococcal meningitis, receiving primary therapy
* Breastfeeding infants whose mothers are receiving or plan to initiate EFV-based highly active antiretroviral therapy (HAART) before the results of the intensive pharmacokinetic (PK) studies are available will be excluded from enrollment in this study due to the potential effect on the infant's EFV PK levels that will be evaluated in the study. More information on this criterion can be found in the protocol.

Ages: 3 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2010-02-10 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Any treatment-related Grade 2B rash or Grade 3 or 4 toxicity requiring permanent discontinuation of efavirenz (EFV) | Measured through Week 24
  Any treatment-related Grade 2B rash or Grade 3 or 4 toxicity requiring permanent discontinuation of efavirenz (EFV)
Death | Measured through Week 24
  Death
A safety event as defined as a Grade 4 life-threatening toxicity or Grade 4 toxicity accompanying a serious adverse event (SAE) (e.g., hospitalization) or death that is judged to be at least possibly related to EFV | Measured through Week 24
  A safety event as defined as a Grade 4 life-threatening toxicity or Grade 4 toxicity accompanying a serious adverse event (SAE) (e.g., hospitalization) or death that is judged to be at least possibly related to EFV
Failure to achieve the area under the curve (AUC) target range despite dose adjustment | Measured through Week 24
  Failure to achieve the area under the curve (AUC) target range despite dose adjustment

SECONDARY OUTCOMES:
A confirmed decrease (less than 1 log) from entry quantitative HIV RNA and RNA greater than 400 copies/mL | Measured at Week 8
  A confirmed decrease (less than 1 log) from entry quantitative HIV RNA and RNA greater than 400 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Bolton, MBBCh, Study Chair — UAB, CIDRZ; Mutsawashe Bwakura-Dangarembizi, MD, Study Chair — Univ. of Zimbabwe, AIDS Research Unit; Ellen Gould Chadwick, MD, Study Chair — Northwestern Univ. Feinberg School of Medicine - Dept. of Peds, Children's Memorial Hosp.
Locations (7):
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- South Africa (4):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Shandukani Research CRS, Johannesburg, Gauteng
  - Durban Paediatric HIV CRS, Durban, KwaZulu-Natal
  - Family Clinical Research Unit (FAM-CRU) CRS, Tygerberg Hills, Western Cape
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Harare Family Care CRS, Harare, Zimbabwe

REFERENCES:
- [Background] ter Heine R, Scherpbier HJ, Crommentuyn KM, Bekker V, Beijnen JH, Kuijpers TW, Huitema AD. A pharmacokinetic and pharmacogenetic study of efavirenz in children: dosing guidelines can result in subtherapeutic concentrations. Antivir Ther. 2008;13(6):779-87. PMID 18839779
- [Background] Kwara A, Lartey M, Sagoe KW, Xexemeku F, Kenu E, Oliver-Commey J, Boima V, Sagoe A, Boamah I, Greenblatt DJ, Court MH. Pharmacokinetics of efavirenz when co-administered with rifampin in TB/HIV co-infected patients: pharmacogenetic effect of CYP2B6 variation. J Clin Pharmacol. 2008 Sep;48(9):1032-40. doi: 10.1177/0091270008321790. PMID 18728241
- [Background] Wintergerst U, Hoffmann F, Jansson A, Notheis G, Huss K, Kurowski M, Burger D. Antiviral efficacy, tolerability and pharmacokinetics of efavirenz in an unselected cohort of HIV-infected children. J Antimicrob Chemother. 2008 Jun;61(6):1336-9. doi: 10.1093/jac/dkn112. Epub 2008 Mar 13. PMID 18343800